CLINICAL TRIAL: NCT06350786
Title: Conditioned Open-label Placebos to Facilitate the Reduction of Opioid Medication (ROM) in Patients With Chronic Non-cancer Pain: a Randomized Controlled Trial
Brief Title: Conditioned Open-label Placebos to Facilitate Opioid Reduction in Patients With Chronic Non-cancer Pain
Acronym: ROM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cosima Locher (Other)
Collaborators: Brown University (Other); University of Basel (Other)
Responsible Party: Sponsor-Investigator, Cosima Locher, Principal Investigator, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROM Study; PZ00P1_201972 (Other Grant/Funding Number: Swiss National Science Foundation)
Record Dates: First submitted 2024-03-14; First posted 2024-04-05 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-02

CONDITIONS: Chronic Non-cancer Pain
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Open-Label Placebo (Experimental): The intervention involves administering "P-Dragees blue Lichtenstein," blue placebo pills devoid of active ingredients. Each pill contains lactose monohydrate; magnesium stearate (Ph. Eur.); microcrystalline cellulose; sucrose; glucose syrup; corn-starch; highly dispersed silicon dioxide; white clay; macrogol glycerol hydroxy stearate (Ph. Eur.); Gum arabic; montanglycol wax; povidone (K 25); talcum; titanium dioxide (E 171); calcium carbonate; macrogol 6000; patent blue V; aluminium salt (E 131).
  Participants will be informed that the pills are placebos and will be instructed to pair them with opioid medication for 7 days. After 7 days until the end of the study they will be instructed to continue to pair their opioid medication with an OLP pill and take additionally placebo pills on the basis of their need.
  An evidence-based rationale will be provided, explaining why the placebo treatment is deemed effective for pain. This rationale will precede the OLP intake procedure.
  Interventions: Other: P-Dragees blue Lichtenstein, Placebo dragees
- Electronic monitoring (EM) control group (Other): EM is a method to objectively measure adherence and serves as the primary intervention component on the basis of which adherence trajectories will be discussed. The participants in the EM control group will receive an evidence-based rational designed to foster positive expectations and will be instructed on the mechanisms of EM.
  The EM control group is structurally equivalent to the OLP group referring to the number and duration of contacts between participants and the study team members as well as to the format of the intervention and the quality of the interaction.
  Interventions: Other: Control group (EM)

INTERVENTIONS:
Other: P-Dragees blue Lichtenstein, Placebo dragees — In the intervention group, open-label placebos are administered within the framework of a mind-body management intervention approach, which in turn is consistent with the biopsychosocial model of pain and with a patient-centred approach. The verbal interaction follows the four discussion points:
  1. Opioids work by telling the body that participants are not experiencing as much pain;
  2. Placebos should be taken every time an opioid is taken which supports the reduction of opioid medication (shown by previous studies);
  3. By pairing the pills together the brain will learn to release chemicals like endorphins that cause pain-relief in response to the placebo, just as it does in response to the opioid;
  4. At a certain point, placebos might provide adequate pain relief, and the participants might need less opioids.
  Arms: Open-Label Placebo
Other: Control group (EM) — In the EM control group, the focus lies on the electronic monitoring (EM) of the opioid intake. The treatment rationale is designed to facilitate the reduction of opioid medication by promoting a positive attitude towards the implementation of the reduction. The verbal interaction follows the four discussion points:
  1. The collection of EM data allows for greater patients' sense of agency over medication treatment;
  2. Tracking of opioid medication use supports the reduction of opioid medication (shown by previous studies);
  3. The EM is a useful tool, and daily recording of opioid medication intake should be done;
  4. At a certain point, EM might provide adequate pain relief, and participants might need less opioids.
  Arms: Electronic monitoring (EM) control group

SUMMARY:
This study aims to evaluate whether the reduction of the daily morphine equivalent dose (MED) in patients with chronic non-cancer pain (CNCP) can be decreased with an open-label placebo (OLP) intervention in comparison to an electronic monitoring (EM) control group. The participants will receive the intervention (OPL or EM) over the duration of six weeks. Diverse psychological and health measures will be assessed with questionnaires over the course of the intervention. Furthermore, evaluation outcomes, qualitative outcomes and safety outcomes will be assessed. It is hypothesized that the OLP-intervention group in comparison to the EM-control group will have a significantly lower consumption of MED over the course of the study. Furthermore, this study aims to evaluate whether the OLP intervention can reduce opioid withdrawal symptoms in comparison to the control group.

DETAILED DESCRIPTION:
CNCP is a major global health problem and is often treated with opiod medication, although risks outweigh the benefits. Therefore, recent studies suggest that an open-label placebo (OLP) treatment, the placebo treatment with full disclosure of being a placebo, has proven to be an effective, clinically relevant, and evidence-based treatment in CNCP syndromes. Furthermore, a new line of research indicated that OLPs have been shown to be feasible for the reduction of active medication in opioid use disorder. In line with the conditioning paradigm, the drug as the unconditioned stimulus is paired with the neutral stimulus of an OLP in a learning phase. Then, the OLP alone becomes a conditioned stimulus.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* ≥ 18 years of age
* German speaking
* Chronic non-cancer pain ≥ 6 months in duration
* Chronic opioid medication for > 3 months
* Oral intake of opioid medication
* Motivation for opioid reduction
* Participants have a primary treating physician who performs the reduction of the opioid medication
* Having access to a computer or tablet with an email-account

Exclusion Criteria:

* Having psychotic symptoms
* Suicidality
* Cognitive impairment to everyday life
* Planned surgery within the next two months
* Known illegal drug or harmful alcohol consumption
* Intolerance of the ingredients of the placebo pill (e.g., lactose, sucrose, corn-starch)
* Serious health problems that make study participation impossible
* Simultaneous participation in other studies with investigational drugs or CNCP specific interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Daily opioid consumption (MED): | Daily measure: starts on day 1 after the first intervention visit (baseline, day 0) after randomization and ends on day 42 at the end of the study.
  Cumulative dose (i.e. total amount) of opioid pain medication consumption based on daily morphine equivalent doses (MED). Data is collected in SEMA3 app.

SECONDARY OUTCOMES:
Subjective opioid withdrawal symptoms | Measured three times: on day 0 at the first intervention visit (baseline), on day 7, and on day 42 at the end of the study.
  Subjective opioid withdrawal will be assessed with the Subjective Opiate Withdrawal Scale (SOWS). The intensity of the withdrawal symptoms is rated by the patient on a scale between 0 (= not at all) and 4 (= extremely), the scores for individual symptoms are added to a total sum score, which can range from 0 to 64. The secondary endpoint will be the subjective opioid withdrawal score at study end (t3).
Pain severity | Measured three times: on day 0 at the first intervention visit (baseline), on day 7, and at the end of the study on day 42.
  Pain severity is assessed using the ICD-11 specifiers or 'extension codes'. The index combines patient-assessed ratings of pain intensity, pain-related distress and pain-related interference. Each of these ratings is assessed on an 11-point NRS rating scale, and these are mapped into the following categories depending on the NRS score: none = NRS 0, mild = NRS 1 - 3, moderate = NRS 4 - 6 and severe = NRS 7 - 10.
Pain disability | Measured three times: on day 0 at the first intervention visit (baseline), on day 7, and at the end of the study on day 42.
  Pain disability is assessed using the pain disability index (PDI) to determine the subjective degree of self-reported impairment caused by the pain problem in everyday life. Seven domains of life are assessed: (1) family and domestic responsibilities, (2) recreation, (3) social activities, (4) occupation, (5) sexual life, (6) self-care and (7) essential activities. The scale ranges from 0 "no impairment" (minimum) - 10 "full impairment" (maximum).
Anxiety | Measured three times: on day 0 at the first intervention visit (baseline), on day 7, and at the end of the study on day 42.
  Anxiety is assessed using the German version of the GAD-7. It is a brief instrument for assessing self-reported generalized anxiety disorder (GAD) symptoms with seven items asking about the main diagnostic criteria of GAD according to the DSM-IV and the ICD-10 criteria. The questions refer to the past two weeks. The scale ranges from "not at all" (minimum); "On some days"; "On more than half of the days"; "almost every day" (maximum).
Depression | Measured three times: on day 0 at the first intervention visit (baseline), on day 7, and at the end of the study on day 42.
  Depression is assessed using Patient Health Questionnaire (PHQ-D) consisting of nine items referring to the past two weeks. The German version of the PHQ was derived from the 'Prime MD Patient Health Questionnaire' and is based on the criteria of the DSM-IV. The scale ranges from "not at all" (minimum); "On some days"; "On more than half of the days"; "almost every day" (maximum).
Pain Opioid Analgesics Beliefs Scale - Cancer | Measured three times: on day 0 at the first intervention visit (baseline), on day 7, and at the end of the study on day 42.
  The POABS-CA in the German version measures pain opioid beliefs based on two components with 10 items and a 5-point Likert scale ranging from 0 ("strongly disagree") to 4 ("strongly agree"). The higher the score, the more negative was the opinion about the use of opioid analgesics for cancer pain, and the stronger was the belief that pain should be endured.
Treatment Expectancy 1 | One-time assessment: measured on day 0 at the first intervention visit (baseline).
  Expectation measures will be measured in analogy to the most relevant outcomes. First, subjectively expected amount (dose) of opioid medication taken will be examined. For this, the following item will be used at the end of the study "How much opioid medication do you think you will be taking at the end of the study?" The item is answered by naming the type of medication, frequency and amount (dose) of medication.
Treatment Expectancy 2 | One-time assessment: measured on day 0 at the first intervention visit (baseline).
  Expectation measures will be measured in analogy to the most relevant outcomes. Second, to measure the expected withdrawal symptoms at the end of the study, items from the SOWS questionnaire will be used, which are expanded with instructions regarding the expectation.
Placebo pill count | Daily measure: starts 1 day after the first intervention visit (baseline, day 0) after randomization and ends on day 42 at the end of the study.
  The intake of placebo pills by the OLP-group will be electronically monitored using survey provided by the app SEMA3. For statistical analysis a ratio will be calculated. A value of the ration close to 1 indicated a more accurate data entry of the placebo pill intake.
Opioid adherence | Daily measure: starts 1 day after the first intervention visit (baseline, day 0) after randomization and ends on day 42 at the end of the study.
  Opioid adherence trajectories will be measured with the app SEMA3 in both groups. In the EM control group, a print of the actual data report from the app (i.e. graph reflecting the pattern of opioid medication intake) will be the basis for the EM-Feedback.

OTHER OUTCOMES:
Rationale credibility | One-time assessment: measured on day 42 at the end of the study.
  The rationale credibility of the OLP intervention will be assessed in the OLP group at study end. The following questions will be assessed: "How credible did you find the explanation of why placebo treatment can work?", "During the study, did you believe that these were placebo tablets that did not contain a pharmacologic agent?", "Did you find the explanation of why the placebo intervention may work helpful?", "How helpful did you find the explanation of why placebo treatment can work?". Answers will be rated on a Likert scale ranging from 0 = Not at all to 4 = Extremely.
Placebo understanding | One-time assessment: measured on day 42 at the end of the study.
  The understanding of placebo will be assessed in both study groups (OLP and control group) at study end using a questionnaire which assesses responders' attitudes regarding non-specific therapies. The first three items of this questionnaire specifically assess the placebo understanding and will be used for this study. The scales differ for the different items.
  Scale question 1: "I have never heard of the term"; "I have heard the term before, but I do not know"; "A placebo is ... (open question)" Scale question 2: "For me the term is rather positive" "For me the term is neutral, neither positive nor negative"; "For me the term is rather negative"; "I do not know" Scale question 3. "Yes, very often"; "Yes, but rarely"; "No"; "I do not know"
  Additionally participants are asked, if their understanding of placebos might have changed across the study. Scale: "Yes, to the positive because ... (open question)"; Yes, to the negative because ... (open question)"; "No"; "I do not know"
Patient Provider Connection | One-time assessment: measured on day 42 at the end of the study.
  The Patient Provider Connection is a subscale of the German version of the Healing Encounters and Attitudes List (HEAL) which can be used independently from the six subscales. The seven items are rated on a five-point Likert scale ranging from "not at all" to "very strong" assessing participants' attitudes towards patient-provider connection as a non-specific treatment effect. The scale ranges from 0 "not at all" (minimum) to "very much" 4 (maximum)
Medication history | Measured two times: on day 0 at the first intervention visit (baseline) and on day 42 at the end of the study.
  Participants' non-opioid medication intake will be assessed by asking the participants about the medication's name, dosage, and reason for intake. Participants will also be asked about the date of prescription.
Primary treating physicians' acceptability of the OLP approach: | One-time assessment, measured before study start: on day -14, prior to the first intervention visit (baseline, day 0).
  Before the start of the study the primary treating physicians will be asked about their acceptability of the OLP approach from patient and physicians point of view. All items will be rated on a five- or seven-point Likert scale.
Primary treating physicians' treatment expectancies | One-time assessment, measured before study start: on day -14, prior to the first intervention visit (baseline, day 0).
  The primary treating physicians will be given the same questionnaire on treatment expectations as the participants. They will be asked about their subjective expectation of their patients' use of opioid medication and their subjective expectation of their patients' withdrawal symptoms at the end of the study. In addition, the primary treating physicians will be asked to assess their patients' motivation to reduce opioid pain medication. Motivation will be assessed with the following questions on a satisfaction ruler ranging from 0 % to 100 %: 1. "How satisfied is your patient currently with his opioid medication?", 2. "How confident are you that your patient can change her/his use of opioid medication?".
Qualitative Outcomes | One-time assessment: measured at the end of the study on day 42.
  The qualitive outcomes will be assessed with an audio recorded semi-structured interviews and will consist of general questions about placebos and core question about the experience of the OLP intervention, acceptability of the OLP approach and prerequisites, ideas and concerns regarding practical OLP implementation.
Additional Symptoms | Measured two times: on day 7 after the first intervention visit (baseline) and on day 42.
  Participants answer three questions regarding additional symptoms that might have occurred since the last visit at the study site.
  The questions are the following:
  * "How have you been since the last visit?" (open answer format)
  * "Did you have certain symptoms?" (yes/no)
  * If the participant answered yes in question 2, a follow up question will be displayed: "Please describe the symptoms you had in detail." (open answer format)

CONTACTS AND LOCATIONS:
Overall Officials: Cosima Locher, PhD, Principal Investigator — USZ
Locations (1):
- University Hospital Zurich, Department of Consultation-Liaison Psychiatry and Psychosomatic Medicine, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (data set and data dictionary)
Supporting Information: Study Protocol
Time Frame: Beginning 6 months after publication
Access Criteria: Researchers with a methodologically sound proposal
URL: https://osf.io

REFERENCES:
- [Background] Buergler S, Sezer D, Gaab J, Locher C. The roles of expectation, comparator, administration route, and population in open-label placebo effects: a network meta-analysis. Sci Rep. 2023 Jul 22;13(1):11827. doi: 10.1038/s41598-023-39123-4. PMID 37481686
- [Background] Belcher AM, Cole TO, Massey E, Billing AS, Wagner M, Wooten W, Epstein DH, Hoag SW, Wickwire EM, Greenblatt AD, Colloca L, Rotrosen J, Magder L, Weintraub E, Wish ED, Kaptchuk TJ. Effectiveness of Conditioned Open-label Placebo With Methadone in Treatment of Opioid Use Disorder: A Randomized Clinical Trial. JAMA Netw Open. 2023 Apr 3;6(4):e237099. doi: 10.1001/jamanetworkopen.2023.7099. PMID 37043203
- [Background] Bernstein MH, Magill M, Weiss AP, Kaptchuk TJ, Blease C, Kirsch I, Rich JD, Becker SJ, Mach S, Beaudoin FL. Are Conditioned Open Placebos Feasible as an Adjunctive Treatment to Opioids? Results from a Single-Group Dose-Extender Pilot Study with Acute Pain Patients. Psychother Psychosom. 2019;88(6):380-382. doi: 10.1159/000503038. Epub 2019 Sep 27. No abstract available. PMID 31563914
- [Background] Estudillo-Guerra MA, Mesia-Toledo I, Schneider JC, Morales-Quezada L. The Use of Conditioning Open-Label Placebo in Opioid Dose Reduction: A Case Report and Literature Review. Front Pain Res (Lausanne). 2021 Jul 12;2:697475. doi: 10.3389/fpain.2021.697475. eCollection 2021. PMID 35295534
- [Background] Flowers KM, Patton ME, Hruschak VJ, Fields KG, Schwartz E, Zeballos J, Kang JD, Edwards RR, Kaptchuk TJ, Schreiber KL. Conditioned open-label placebo for opioid reduction after spine surgery: a randomized controlled trial. Pain. 2021 Jun 1;162(6):1828-1839. doi: 10.1097/j.pain.0000000000002185. PMID 33449503
- [Background] Morales-Quezada L, Mesia-Toledo I, Estudillo-Guerra A, O'Connor KC, Schneider JC, Sohn DJ, Crandell DM, Kaptchuk T, Zafonte R. Conditioning open-label placebo: a pilot pharmacobehavioral approach for opioid dose reduction and pain control. Pain Rep. 2020 Jul 20;5(4):e828. doi: 10.1097/PR9.0000000000000828. eCollection 2020 Jul-Aug. PMID 32766465
- [Background] Sezer D, de Leeuw M, Netzer C, Dieterle M, Meyer A, Buergler S, Locher C, Ruppen W, Gaab J, Schneider T. Open-Label Placebo Treatment for Acute Postoperative Pain (OLP-POP Study): Study Protocol of a Randomized Controlled Trial. Front Med (Lausanne). 2021 Nov 5;8:687398. doi: 10.3389/fmed.2021.687398. eCollection 2021. PMID 34805194
- [Derived] Carratta K, Bodonyi K, Frey Nascimento A, Friis D, von Kanel R, Bircher L, Koechlin H, Bernstein M, Streitberger K, Arnet I, Roth AJ, Ronel J, Olliges E, Locher C. Conditioned open-label placebos to facilitate opioid reduction in patients with chronic non-cancer pain: study protocol of a randomised controlled trial. BMJ Open. 2025 May 24;15(5):e098253. doi: 10.1136/bmjopen-2024-098253. PMID 40413049